CLINICAL TRIAL: NCT00396838
Title: Cardiac Autonomic Reactivity and Behavioral Response to Pain in Full-Term Neonates
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: 1909CTIL
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background: Heel lancing is a routine procedure for the diagnosis of phenylketonuria in infants. Despite the short- and long-term adverse effects of pain, there are no guidelines for the reduction of such pain. Previous studies evaluated different treatment modalities; however, in most of them, pain response was assessed by subjective measures.

Aims of study: 1. To characterize the pain response of infants by using a computerized analysis of the ECG. 2. To compare six different methods of pain reduction during heel lancing in newborns.

Methods: The time, geometric and frequency domains of the infants' ECG will be computed during heel lancing. 150 healthy full-term infants will be evaluated in six treatment groups: breastfeeding, bottle feeding, skin-to-skin contact, lying on a table without anything, lying with a pacifier and lying while getting a glucose solution. The differences in pain response to these six treatment modalities will be assessed and compared to the infants' length of cry, and scoring of the infants' behavioral response.

ELIGIBILITY:
Inclusion Criteria:

* normal full-term newborns (>38 weeks)
* Apgar score >=8 at five minutes after delivery.

Exclusion Criteria:

* congenital anomalies
* medical complications
* need for oxygen administration

Ages: 48 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Weissman, MD, Study Director — Rambam MC
Locations (1):
- Rambam MC, Haifa, Israel

REFERENCES:
- [Derived] Weissman A, Aranovitch M, Blazer S, Zimmer EZ. Heel-lancing in newborns: behavioral and spectral analysis assessment of pain control methods. Pediatrics. 2009 Nov;124(5):e921-6. doi: 10.1542/peds.2009-0598. Epub 2009 Oct 19. PMID 19841119